CLINICAL TRIAL: NCT04708132
Title: Prosthetic Maintenance and Peri- Implant Tissues Conditions of Fixed Screw- Retained Implant Prosthesis Versus Implant-Retained Ball Overdentures: A Randomized Clinical Trial
Brief Title: Maintenance and Tissues Conditions of Fixed Screw-Retained Implant Prosthesis Versus Implant-Retained Ball Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Ragheb, principal invistigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KD/02/20
Record Dates: First submitted 2021-01-06; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Prosthesis and Implant Dentistry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- screw retained restorations (Active Comparator)
  Interventions: Procedure: Screw retained restoration
- implant-retained ball overdentures (Other)
  Interventions: Procedure: implant-retained ball overdentures

INTERVENTIONS:
Procedure: Screw retained restoration — Hybrid prosthesis
  Arms: screw retained restorations
Procedure: implant-retained ball overdentures — Removable prosthesis
  Arms: implant-retained ball overdentures

SUMMARY:
The aim of this study was to compare the prosthetic maintenance requirements between implant-retained ball overdentures versus fixed screw- retained implant prosthesis. Clinical and radiographic changes in peri-implant tissue with using PGE2 as a PICF biomarker were also evaluated. Selected patients had been divided into two groups:

1. Group (I): twenty seven patients had received implant-Supported ball over dentures.
2. Group (II): twenty-seven patients had received screw retained restorations Interventions and study procedures

Surgical and prosthetic procedures:

Surgical Procedures A radiopaque radiographic stent was formed and was positioned in the patient's mouth during cone beam scanning. Four implants were planned with two virtual replicas, in the place of the lateral incisor and the second premolar.

The stent was fabricated. After the healing period of four months finished, the patients were recalled and the super structure was fabricated according to the type of restoration Follow-up During the 12 months follow-up period, prosthodontic complications were recorded and calculated.

Postoperative care Along with a conventional oral hygiene assessment and functional checkup, follow up visits were scheduled every 6 months and up to 12 months total follow up period.

Clinical soft tissue measurements which include plaque index (PI), gingival index (GI), and PPD were measured at the mid-facial, mid-lingual, mid-mesial, and mid-distal aspects of each fixture using a graduated plastic probe to the nearest 0.5 mm. These clinical measurements were recorded after prosthesis delivery, 6 and 12 months postoperatively. The peri-implant marginal bone loss (MBL) was assessed radiographically after prosthesis delivery, 6 and 12 months postoperatively.

• Collection of peri-implant crevicular fluid (PICF) samples: PICF was collected.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients have Angle Class I maxilla-mandibular relationship.
* Age range between 40 and 70.
* Maxillary and mandibular ridges with no history of fresh extraction.
* Sufficient bone volume to house four implants in each arch.
* Sufficient zone of keratinized attached mucosa >5mm over the crest of the upper and lower ridges.

Exclusion Criteria:

* the patients have a past history of head and neck radiation
* previous ridge augmentation or grafting
* Lack of any systemic diseases that could affect osseointegration of implants as uncontrolled diabetes , hypertension , and osteoporosis
* Heavy smokers who exceeding 20 cigarette/ day
* para-functional habits for example bruxism or clenching.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Rate of prosthetic complications | 12 months

SECONDARY OUTCOMES:
changes in peri-implant tissue with using PGE2 as a PICF biomarker | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan Ragheb, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry , Kafrelshiekh university, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt